CLINICAL TRIAL: NCT02860221
Title: Intravenous Versus Topical Administration of Low Dose Epinephrine Plus Combined Administration of Intravenous and Topical Tranexamic Acid (TXA)for Primary Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Liu Yang, Professor, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Knee blood
Record Dates: First submitted 2016-07-28; First posted 2016-08-09 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Blood Loss
Keywords: Arthroplasty, Replacement, Knee; Epinephrine; Tranexamic acid
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intravenous epinephrine (Experimental): Intravenous (IV) low dose epinephrine
  Interventions: Drug: Tranexamic acid (TXA); Drug: Epinephrine
- Topical epinephrine (Experimental): Topical epinephrine
  Interventions: Drug: Tranexamic acid (TXA); Drug: Epinephrine
- Control (Active Comparator): No epinephrine
  Interventions: Drug: Tranexamic acid (TXA)

INTERVENTIONS:
Drug: Tranexamic acid (TXA) — IV and topical administration
Drug: Epinephrine
  Arms: Intravenous epinephrine; Topical epinephrine

SUMMARY:
The purpose of this study is to compare the blood loss of intravenous and topical administration of low dose epinephrine plus combined administration of intravenous and topical tranexamic acid for primary total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* All patients between the ages of 20 and 75 who were diagnosed with osteoarthritis of the knee and scheduled for an elective primary total knee arthroplasty and those who were willing and able to return for follow-up over at least a 6-month postoperative period

Exclusion Criteria:

* Acute coronary syndrome < 6 months
* Glaucoma,pheochromocytoma, thyrotoxicosis, digoxin intoxication, serum potassium < 3.0 mmol, alcohol abuse, premenopausal women
* Current treatment with adenosine diphosphate (ADP) receptor antagonists, Factor Xa or thrombin inhibitors,heparin (excluding Low Molecular Weight Heparin (LMWH) for perioperative thromboprophylaxis), tricyclic antidepressants, or monoamine oxidase（MAO) or Catechol-O-methyltransferase (COMT) inhibitors
* Patients with history of thromboembolic disease, bleeding disorder
* Patients with history of renal impairment, cardiovascular diseases (previous myocardial infarction, atrial fibrillation) or cerebrovascular conditions (previous stroke or peripheral vascular surgery)
* Allergy to TXA

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-07 (Estimated); Study Completion 2017-07

PRIMARY OUTCOMES:
Total blood loss on the post-operative day 1 | 1 day post-operation

SECONDARY OUTCOMES:
Haemoglobin (Hb) | 7 day
  g/L
Hematocrit (Hct) | 7 day
  Percentage
Blood platelet count (PLT) | 7 day
Post-operation Hospital for special surgery score (HSS) | 3 months
  Scoring
Preoperative and post-operation range of motion (ROM) of operated knee joint (degree) | Through study completion, an average of 3 months
  There is only one Unit of Measure for ROM, it is degree
Length of hospital stay (days) | 3 months
  Days
Number of patients with infection | 3 months
  Post-operatively
Number of deep vein thrombosis (DVT) cases | 1 month
  Post-operatively
Number of pulmonary embolism (PE) cases | 1 month
  Post-operatively
Intraoperative blood loss | 3 hours
  Post-operatively
Intravenous fluid administration on the operation day | 1 day
  Milliliter
Total blood loss on the post-operative day 3 | 3 day post-operation
  Milliliter
Reaction time (R-time) | 24 hours
Rate of thrombus formation (K time) | 24 hours
Maximum amplitude (MA) | 24 hours
Rate of thrombus formation (α-angle) | 24 hours
Lysis rate at 30 min (LY30) | 24 hours
Coagulation index (CI) | 24 hours
Interleukin(IL)-1β | 24 hours
Interleukin(IL)-6 | 24 hours
Interleukin(IL)-8 | 24 hours
Tumor necrosis factor (TNF)-α | 24 hours
C-reactive protein (CRP) | 24 hours
Interleukin(IL)-10 | 24 hours
Wound score | 14 day
Blood transfusion rate | 7 day
Blood transfusion volume (mL) | 7 day

CONTACTS AND LOCATIONS:
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No